CLINICAL TRIAL: NCT02494947
Title: Physical Activity and Lipid Content of Coronary Artery Atheromatous Plaques: a Randomised Trial Using Novel Intracoronary Imaging Techniques
Brief Title: Coronary Disease and the Effect of High-intensity Interval Training
Acronym: CENIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015/210
Record Dates: First submitted 2015-07-06; First posted 2015-07-10 (Estimated); Last update posted 2019-08-26 (Actual); Status verified 2019-08

CONDITIONS: Coronary Disease
Keywords: Coronary Angiography; Exercise
MeSH Terms: conditions — Coronary Disease; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- interval training (Experimental): high intensity interval-based aerobic exercise
  Interventions: Behavioral: high intensity interval-based aerobic exercise; Other: Usual care
- controls (Other): usual care
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: high intensity interval-based aerobic exercise — Interval exercises done 3 times weekly during 6 months according to standard procedures at the Department of Circulation and Medical Imaging.
  Arms: interval training
Other: Usual care

SUMMARY:
The primary purpose of this study is to investigate if systematic, high intensity, interval-based aerobic exercise training results in regression of lipid content of atherosclerotic coronary artery plaques, and in reduction of plaque burden in patients with stable coronary heart disease. Composition and morphologic characteristics of plaques will be studied by intra-coronary near-infrared spectroscopy (NIRS) and intravascular ultrasound (IVUS) in patients undergoing percutaneous coronary intervention.

ELIGIBILITY:
Inclusion Criteria:

* stable coronary artery disease
* will undergo cardiac catheterization
* will be treated with percutaneous coronary intervention (PCI)
* signed written informed consent
* able to execute the intervention

Exclusion Criteria:

* earlier bypass surgery
* known inflammatory disease other than atherosclerosis
* planned surgery within 4 months
* included in another randomized controlled study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
lipid content of atherosclerotic coronary artery plaques | 6 months
  Lipid core burden index (LCBI) measured by intracoronary near-infrared spectroscopy

CONTACTS AND LOCATIONS:
Overall Officials: Rune Wiseth, phd prof, Study Director — Norwegian University of Science and Technology
Locations (1):
- St Olavs Hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Vesterbekkmo EK, Madssen E, Aamot Aksetoy IL, Follestad T, Nilsen HO, Hegbom K, Wisloff U, Wiseth R. CENIT (Impact of Cardiac Exercise Training on Lipid Content in Coronary Atheromatous Plaques Evaluated by Near-Infrared Spectroscopy): A Randomized Trial. J Am Heart Assoc. 2022 May 17;11(10):e024705. doi: 10.1161/JAHA.121.024705. Epub 2022 May 16. PMID 35574968